CLINICAL TRIAL: NCT05380154
Title: Phase 3 Clinical Study of Efficacy and Safety Assessment; Multi-center, Randomized, Blind, and Parallel Control; and Positive Control of Botulax® Injection and BOTOX® for Improvement of Moderate to Severe Glabellar Wrinkles
Brief Title: Efficacy and Safety Assessment of Botulax® and BOTOX® for Improvement of Glabellar Lines.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hugel (Industry)
Collaborators: Sihuan Pharmaceutical Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Botulax-3001
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-04

CONDITIONS: Glabellar Lines
Keywords: botulinum toxin type A; Glabellar lines; wrinkles
MeSH Terms: interventions — Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators (investigator, evaluator at each institution, photographer, Independent Evaluation Committee, etc.), except for the injection mixing officer, employees of the sponsor, and test subjects are blinded during the test. Each institution appoints an independent injection formulation officer and prohibits interchange with the drug substance test group to make sure that the blinded method of the test is performed accurately
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Botulinum Toxin A type for injection (Botulax®)
  Interventions: Drug: Botulinum Toxin A type for injection (Botulax®)
- control group (Active Comparator): Botulinum Toxin A type for injection (BOTOX®, Bao Tuo Shi®)
  Interventions: Drug: Botulinum Toxin A type for injection (BOTOX®, Bao Tuo Shi®)

INTERVENTIONS:
Drug: Botulinum Toxin A type for injection (Botulax®) — Person in charge of dilution uses 0.9% sodium chloride injection solution to formulate the drug substance into 4U/0.1mL composite solution, and the investigator injects it into the test subjects
  Arms: Test group
Drug: Botulinum Toxin A type for injection (BOTOX®, Bao Tuo Shi®) — Person in charge of dilution uses 0.9% sodium chloride injection solution to formulate the drug substance into 4U/0.1mL composite solution, and the investigator injects it into the test subjects.
  Arms: control group

SUMMARY:
This study is a phase 3 clinical trial of multi-center, random, blinded*, parallel control, and positive control to evaluate the efficacy and safety of Botulax® Injection compared to BOTOX® for improving moderate to severe glabellar wrinkles.

DETAILED DESCRIPTION:
The case test of 500 qualified test subjects was conducted in 13 institutions nationwide in China. Those who meet all selection criteria and do not meet any of the exclusion criteria are selected as suitable test subjects. The selected test subjects are blinded and divided into the Botulax test group or the BOTOX test group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 65 years (inclusive), no gender preference
2. The evaluator at each institution assesses the severity level of glabellar wrinkles at the site in the field when the test subject frowns as much as possible according to the 4-point photographic evaluation table and classifies the subjects with a rating of ≥ 2 (medium or severe).
3. Persons who can follow the test well, fully understand the clinical trial, rationally foresee the cost-effectiveness of injection, and adhere to the study procedure until the end of the clinical trial are selected.
4. The test subjects fully understand the test requirements and voluntarily sign the consent form.

Exclusion Criteria:

1. Subjects who have a history of oversensitivity to the Botulinum Toxin A type, Botulinum Toxin B type, or other control groups of the tested drug substance.
2. Subjects with clear scars, infections, a carcinogenic or cancerous metastatic lesion on the upper part of the face and/or unrecovered wounds on the face.
3. Subjects with skin disease, such as dermatitis and acne, or scar on the face, which the investigator judges can affect the evaluation of treatment effectiveness or safety of the test subject.
4. Subjects who took anticoagulant drugs (e.g., aspirin, nonsteroidal anti-inflammatory drugs, clopidogrel, warfarin, etc.) within two weeks prior to selection; the test subjects who are menstruating can avoid it by delaying the injection of studied products as needed.
5. Subjects who took drugs with muscle relaxation effects (e.g., muscle relaxants, Curare-like substances, anticholinergic drugs, spectinomycin hydrochloride, aminoglycoside-based drugs, polypeptide antibiotics, tetracycline, lincomycin-based drugs, anticholinergics, benzodiazepines and similar drugs, or benzamide drugs) within 4 weeks prior to selection, anticholinergics, benzodiazepines and similar drugs, or benzamide drugs) or are foreseen to use the above drugs during the study period (for 16 weeks after the injection treatment).
6. Subjects who have used external medications (e.g., glucocorticoids or tretinoin ointment) on the upper part of the face within 4 weeks prior to the selection or are foreseen to use the drug on the upper part of the face during the study period (for 16 weeks after the injection treatment).
7. Subjects who have a history of injecting drugs similar to the study drug within 6 months prior to selection or are foreseen to use during the study period (Botulinum Toxin A type or Botulinum Toxin B type).
8. Subjects who have undergone eye shape correction, laser skin transplantation, skin surgery, IPL, frequency surgery, dermabrasion, chemical dermabrasion, or other laser resolution and nonresolution surgery within 6 months prior to selection or are foreseen to do so during the study period.
9. Subjects who have had injected hyaluronic acid in the upper part of their face within 12 months prior to selection or plan to do it.
10. Subjects who have a history of surgery to remove wrinkles on the face above the eyes or a permanent filling injection.
11. Subjects who plan to undergo a wrinkle removal surgery on their face during the study period, an injection filling of soft tissue for wrinkle removal, or other facial plastic surgeries.
12. Subjects whom the investigator judges to be unsuitable to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Responder rate of improvement in glabellar lines with Physician's rating of line severity | Week 4
  The rate of test subjects receiving 0 or 1 point by the institution evaluator who assesses the glabellar wrinkles (at maximum frown) at the site in week 4.

SECONDARY OUTCOMES:
Responder rate of improvement in glabellar lines with Physician's rating of line severity | weeks 1, 8, 12, and 16 after the treatment
  The rate of test subjects receiving 0 or 1 point by the institution evaluator who assesses the glabellar wrinkles (at maximum frown)at the site in weeks 1, 8, 12, and 16 after the treatment
Responder rate of improvement in glabellar lines at rest with Physician's assessment of severity | weeks 1, 4, 8, 12, and 16 after the treatment
  The rate of test subjects receiving 0 or 1 point by the institution evaluator who assesses the glabellar wrinkles (when at rest) at the site in weeks 1, 4, 8, 12, and 16 after the treatment
Responder rate of improvement in glabellar lines at maximum frown with investigator's photo assessment | weeks 1, 4, 8, 12, and 16 after the treatment
  The rate of test subjects receiving 0 or 1 point by the Independent Evaluation Committee based on the photo of the glabellar wrinkles (at maximum frown) in weeks 1, 4, 8, 12, and 16 after the treatment
Responder rate of improvement in glabellar lines at rest with investigator's photo assessment | weeks 1, 4, 8, 12, and 16 after the treatment
  The rate of test subjects receiving 0 or 1 point by the Independent Evaluation Committee based on the photo of the glabellar wrinkles (when at rest) in weeks 1, 4, 8, 12, and 16 after the treatment
Responder rate of improvement in glabellar lines with Subject's improvement assessment | weeks 1, 4, 8, 12, and 16 after the treatment
  The rate of test subjects who self-assess that the treatment is effective (by giving a score of "+2" or higher) in weeks 1, 4, 8, 12, and 16 after the treatment
Subject's satisfaction rate | weeks 1, 4, 8, 12, and 16 after the treatment
  The rate of test subjects who are satisfied with the treatment effect (test subject's satisfaction rating of 6 - 7) in weeks 1, 4, 8, 12, and 16 after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hugel Inc., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No